CLINICAL TRIAL: NCT00994968
Title: Neoadjuvant Doxorubicin and Cyclophosphamide Followed by Docetaxel and S-1 in Breast Cancer
Brief Title: Doxorubicin Hydrochloride, Cyclophosphamide, Docetaxel, and S-1 Before Surgery in Treating Women With Stage II or Stage III Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000650694; YONSEI-YCC-BR09-01
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage III breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: tegafur-gimeracil-oteracil potassium
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride, cyclophosphamide, docetaxel, and S-1, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying giving doxorubicin hydrochloride together with cyclophosphamide, docetaxel, and S-1 before surgery in treating women with stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of pathologic complete response in women with previously untreated stage II or III breast cancer treated with neoadjuvant doxorubicin hydrochloride and cyclophosphamide followed by docetaxel and S1.

Secondary

* Determine the safety and tolerability of this regimen in these patients.
* Determine the rate of overall radiologic response in these patients.
* Determine the rate of breast-conserving procedures in these patients.
* Determine the disease-free survival of these patients.
* Investigate the relevant pharmacogenomics and biomarker(s) which will be useful to predict any responses to the anticancer treatments.

OUTLINE: Patients receive neoadjuvant doxorubicin hydrochloride IV and cyclophosphamide IV on day 1. Treatment repeats every 3 weeks for up to 4 courses. Patients then receive docetaxel IV over 1 hour on day 1 and oral S-1 on days 1-14. Treatment repeats every 3 weeks for 4 courses. Two to four weeks later, patients undergo surgery to remove the tumor (either breast-conserving procedures or mastectomy). Patients may then undergo radiotherapy and receive endocrine therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive primary breast cancer

  * Clinical (radiologic) stage II or III disease
  * No T4d disease
  * No inflammatory breast cancer
* ErbB2-negative disease OR patient cannot receive trastuzumab treatment

  * ErbB2-positive disease defined as either immunohistochemistry 3+, or FISH- or CISH-positive; immunohistochemistry 2+ is to be determined according to FISH or CISH results

PATIENT CHARACTERISTICS:

* Mobile
* ECOG performance status 0-1
* Normal cardiac function (LVEF > 50%)
* Hemoglobin ≥ 10.0 g/dL
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 10 x 10^4/μL
* Creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance ≥ 50 mL/min
* Total bilirubin ≤ 1.5 times ULN
* AST/ALT ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow tablet whole with water
* No prior motor or sensory neurotoxicity CTCAE ≥ grade 2
* No other serious disease or medical condition
* No uncontrolled or serious cardiovascular disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class III or IV heart failure
  * Uncontrolled angina pectoris
  * Clinically significant pericardial disease
  * Cardiac amyloidosis
* No history of symptomatic or therapy-requiring cardiac arrhythmia CTCAE grade 3 (e.g., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, uncontrolled atrial fibrillation)
* No asymptomatic sustained ventricular tachycardia
* History of atrial fibrillation or cardiac arrhythmia controlled by medication allowed
* No uncontrolled infection, unstable peptic ulcer, uncontrolled diabetes, or any other contraindication to corticosteroid administration
* No history of infection or any other serious medical event which may cause any functional injury in the affected patient and consequently, interfere with continuing the study treatment
* No history of hypersensitivity to taxanes, fluorouracil, or S-1
* No significant gastrointestinal malfunction that will affect S-1 absorption
* No history of other cancer within the past 5 years except properly treated carcinoma in situ of the uterine cervix or basal cell or squamous cell carcinoma of the skin
* No severe psychological or neurological disorder or dementia that would preclude understanding of the informed consent
* No psychological, social, family, or geographical condition, or difficult circumstance that would preclude follow-up or compliance with the protocol

PRIOR CONCURRENT THERAPY:

* No prior systemic treatment for this cancer (e.g., radiotherapy, chemotherapy, hormone therapy, or biological therapy)
* No prior preoperative topical treatments (e.g., incomplete surgery or radiotherapy) for this cancer
* No concurrent drug(s) that may potentially cause changes in the pharmacological activity of S-1 formulation, including any of the following:

  * Allopurinol
  * Phenytoin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2009-07

PRIMARY OUTCOMES:
Rate of pathologic complete response

SECONDARY OUTCOMES:
Safety and tolerability
Rate of overall radiologic response
Rate of breast-conserving procedure
Disease-free survival
Relevant pharmacogenomics and biomarker(s) which may be useful to predict any responses to the anticancer treatments

CONTACTS AND LOCATIONS:
Overall Officials: Joo Hyuk Sohn, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Moon YW, Lee S, Park BW, Kim EK, Kim SI, Koo JS, Park S, Kim MJ, Chung HC, Kim JH, Sohn J. S-1 combined with docetaxel following doxorubicin plus cyclophosphamide as neoadjuvant therapy in breast cancer: phase II trial. BMC Cancer. 2013 Dec 6;13:583. doi: 10.1186/1471-2407-13-583. PMID 24314307